CLINICAL TRIAL: NCT04202081
Title: Voices From the Black Community: Beliefs and Attitudes on Participating in Research Studies for Chronic Hepatitis C
Brief Title: Voices From the Black Community: Hepatitis C Research Participation
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 18-0662
Record Dates: First submitted 2019-12-11; First posted 2019-12-17 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Hepatitis C, Chronic
Keywords: patient-reported outcomes; observational; HCV; Hepatitis C; Chronic Liver Disease; Liver Disease; Research; Participation
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Liver Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a one-time cross-sectional survey study of approximately 200 self-identified black or African-American patients who have had chronic hepatitis C viral infection (HCV) that will evaluate patients' willingness to participate (WTP) in health/medical research related to HCV and attitudinal factors that might be associated with WTP, such as benefits and barriers to research participation, mistrust of physicians/researchers, health literacy, and knowledge of health/research studies.

DETAILED DESCRIPTION:
Chronic hepatitis C viral (HCV) infection is three times more prevalent in the African American/black (AA) population than in white patients in the U.S.; yet minorities are woefully under-represented in HCV research, particularly in Phase III drug registration trials. A recent systematic review of randomized controlled clinical trials (RCT) of HCV treatments with interferon-based treatments from 2000 to 2011 found that the proportion of African-American patients in RCTs ranged from 0% - 11%. Despite significant increases in efficacy and reductions in adverse events associated with the new direct acting antiviral (DAA) regimens, the proportion of black patients enrolled in Phase II-III DAA registration trials has not increased dramatically and generally ranges from 1%-18%. Because participation rates in medical research do not fully represent the overall U.S. population or prevalence rates among various subgroups, the Food and Drug Administration (FDA) has mandated pharmaceutical companies to improve demographic subgroups included in clinical trials, to identify barriers to subgroup enrollment in clinical trials, and to employ strategies to encourage greater participation.

Enrolling more diverse patients in medical research, especially racial minorities, is a ubiquitous dilemma that has received a fair amount of scientific attention in the last 10 years. This research has found an important role for the perceptions and attitudes that people have about participating in clinical research. Negative perceptions serve as barriers to enrollment in clinical research, while positive attitudes are facilitators of research participation. Additionally, knowledge gaps, patient-provider communication, health literacy, and mistrust of research and scientists are a few of the commonly reported barriers to participation among minority patients. To our knowledge, no study has been undertaken with black patients with HCV to understand their specific attitudes and perspectives related to participation in HCV-related health or medical research. This information is a prerequisite to developing effective approaches to increasing participation of the black community in HCV-related health or medical research.

Two hundred Black patients will be recruited. Patients who participated in The Patient-Reported Outcomes Project of HCV-TARGET ("PROP UP TARGET") study will be invited to participate. Patients will also be recruited from liver clinics at one medical center. Patients will respond to several survey questions over the phone or in person related to WTP and attitudinal factors related to clinical research.

Participant responses and characteristics will be summarized using graphical and tabular descriptive statistical methods such as sample means, percentiles, frequencies, proportions and standard deviations. All statistical estimates will be reported with confidence intervals.

ELIGIBILITY:
Inclusion Criteria

* Previous enrollment in the Patient-Reported Outcomes Project (PROP UP) or recruited from HCV Liver Clinics at the University of North Carolina.
* Self-identified as African-American or Black during the PROP UP study or in-person
* Provide written or verbal permission to be contacted about future research studies

Exclusion Criteria

* Express unwillingness to be contacted about future studies
* Withdrew from PROP UP post-enrollment (eg. death, patient withdrawal)
* Unwilling or unable to provide verbal consent
* Identifies during the phone survey or in-person that he/she is not African-American or Black

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who self-identify as black or African-American and have been infected with chronic hepatitis C viral (HCV) infection. Patients will be recruited from the Patient-Reported Outcomes Project (PROP UP) observational study (11 U.S. liver centers) and from a tertiary care liver HCV clinic.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-06-19 (Actual)

PRIMARY OUTCOMES:
Overall Willingness to Participate (WTP) Mean Score | through study completion, an average of 1 day
  Overall Willingness to Participate Scale (WTP): WTP in research studies was evaluated using 13 items to assess WTP in different types of health/medical research studies. Responses were based on a five-point Likert scale from 1 (not at all willing) to 5 (very willing), with 3 connoting "unsure/neutral." The overall WTP score will be calculated for each participant by taking the mean of the 13 items. Higher scores indicate higher WTP.

SECONDARY OUTCOMES:
Perceived Benefits/Advantages of Participating in Health/Medical Research Mean Score | through study completion, an average of 1 day
  Perceived Benefits Scale: Patients respond to 16 items regarding perceived benefits or advantages of research participation. Each item is rated on a 5 point likert scale: 1=strongly disagree, 2=disagree, 3=unsure, 4=agree, 5=strongly agree. The average of all items will be used to create the total mean benefit score. Higher scores indicate higher Perceived Benefits.
Perceived Barriers/Disadvantages of Participating in Health/Medical Research Mean Score | through study completion, an average of 1 day
  Perceived Barriers Scale: Patients respond to 12 items regarding barriers or disadvantages of research participation. Each item is rated on a 5 point likert scale: 1=strongly disagree, 2=disagree, 3=unsure, 4=agree, 5=strongly agree. The average of all items will be used to create the total mean barrier score. Higher scores indicate higher Perceived Barriers.
Perceived Trust in Doctors Mean Score | through study completion, an average of 1 day
  Trust in Doctors Scale: Patients respond to 12 items regarding their trust or mistrust in their medical providers. Each item is rated on a 5 point likert scale: 1=strongly disagree, 2=disagree, 3=unsure, 4=agree, 5=strongly agree. Negative items were reverse scored. The average of all items will be used to create the total mean trust score. Higher scores indicate higher Perceived Trust.
Perceived Health Literacy Mean Score | through study completion, an average of 1 day
  Perceived Health Literacy Scale: Three items assessed the health literacy of participants with a five-point response scale: 1 (Never), 2 (Rarely), 3 (Sometimes), 4 (Often), 5 (Always). Participants were asked (a) how frequently they asked others to help them read medical materials, (b) if they felt uncomfortable filling out medical forms, and (c) if they did not understand their medical condition due to difficulty reading medical materials. The average of all items will be used to create the total mean health literacy score. Lower scores indicate higher Perceived Health Literacy.
Subjective Knowledge of Health/Medical Research Mean Score | through study completion, an average of 1 day
  Subjective Knowledge Scale: Participants were asked how well they felt they understood what health/medical research involved. This was assessed on a five-point response scale: 1 (Not at all), 2 (Not too well), 3 (Somewhat well), 4 (Pretty well), 5 (Very well). The average of all items will be used to create the total mean subjective knowledge score. Higher scores indicate higher subjective knowledge.
Objective Knowledge of Health/Medical Research Mean Score | through study completion, an average of 1 day
  Objective Knowledge Scale: Knowledge of clinical trials was measured with 10 true/false questions about aspects of clinical trials. The proportion of correct responses per patient will be recorded. Higher proportion indicates higher objective knowledge.

OTHER OUTCOMES:
Proportion of Participant Recommendations for Strategies | through study completion, an average of 1 day
  Open-ended qualitative question to solicit participants' recommendations for strategies to enhance racial diversity in HCV-related research studies. Responses will be categorized into different recommendation strategies and proportion of patients who listed a strategy in that category will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Donna M Evon, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan at this time to make individual participant data available to other researchers.